CLINICAL TRIAL: NCT05977621
Title: Acquisition of Trans-Rectal Ultrasound [TRUS] Images of the Female Pelvis for Real-Time MRI-US Fusion Based Needle Tracking for Image-Guided Brachytherapy: A Pre-feasibility Study
Brief Title: Trans-Rectal Ultrasound of the Female Pelvis for Real-Time MRI-US Fusion Based Needle Tracking
Acronym: (TRUS)
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: Eigen (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00113768
Record Dates: First submitted 2023-07-28; First posted 2023-08-04 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Uterine Cancer
MeSH Terms: conditions — Uterine Neoplasms | interventions — Ultrasound, High-Intensity Focused, Transrectal

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intact anatomy: Patients with intact anatomy (uterus and cervix)
  Interventions: Other: Transrectal ultrasound (TRUS)
- Post-hysterectomy: Post-hysterectomy patients (vaginal cuff) who are planned to receive brachytherapy
  Interventions: Other: Transrectal ultrasound (TRUS)

INTERVENTIONS:
Other: Transrectal ultrasound (TRUS) — Transrectal ultrasound (TRUS) images of the female pelvis

SUMMARY:
The purpose of this study is to utilize transrectal ultrasound (TRUS) images of the intact and post-hysterectomy female pelvis in order to provide feasibility information for a Magnetic Resonance Imaging (MRI)-TRUS fusion based 3D needle navigation system for use in image guided brachytherapy. The fusion and needle guidance will be performed using Eigen Health's navigation system that currently provides targeted MR/Ultrasound fusion based prostate biopsies utilizing a proprietary 3D semi-robotic navigation system.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven invasive primary squamous, adenosquamous, or adenocarcinoma of the uterine cervix, (recurrent or medically inoperable) uterine adenocarcinoma.
* Treatment plan must include curative-intent definitive radiation that includes brachytherapy treatments with or without concurrent chemotherapy
* Adults ≥ 18 years of age
* ECOG Performance Status 0-2

Exclusion Criteria:

* Patients with active rectal bleeding or rectal ulcer

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Patients who are undergoing brachytherapy as part of the standard plan for their gynecologic cancer diagnosis (defined above) will be our target population. Only women will be eligible for this study. Women of all races/ethnicities will be eligible, and accrual is expected to reflect the population of patients seen in the Duke Radiation Oncology Clinic.
Sampling Method: Non-Probability Sample
Enrollment: 8 (Actual)
Dates: Start 2024-02-07 (Actual); Primary Completion 2025-12-11 (Actual); Study Completion 2025-12-11 (Actual)

PRIMARY OUTCOMES:
Number of patients whose MRI and ultrasound images are fused | up to 5 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Dianda Ayala-Peacock, MD, Principal Investigator — Duke University Health System (DUHS)
Locations (1):
- Duke Cancer Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No